CLINICAL TRIAL: NCT04274296
Title: Advisory Lead ARDS Respirator Management
Acronym: ALARM
Status: Completed | Type: Observational
Sponsor: Mathias Maleczek (Other)
Collaborators: Philips Austria GmbH (Unknown); Medical University of Vienna (Other)
Responsible Party: Sponsor-Investigator, Mathias Maleczek, Registrar, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: ALARM
Record Dates: First submitted 2019-09-30; First posted 2020-02-18 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Control: Control-cohort in which no change in care is needed
- Advisory: Cohort in which advisory is activated
  Interventions: Device: Activation of Advisory

INTERVENTIONS:
Device: Activation of Advisory — Advisory is activated which will show if driving pressure is greater or equal 15
  Groups: Advisory

SUMMARY:
A advisory will be activated in the ICUs patient data management system. The trial will be conducted as observational cohort trial. During the first six month all patients with a LIPS ≥ 4 will be included in the control group. No change of care is needed. In a second phase during the next six months, all patients with a LIPS ≥ 4 will be included into the advisory group where advisories will be shown in the patient data management system.

To create this advisory, a clinical advisory rule is executed every 4 hours and the appropriate advisory text is calculated. If the defined threshold values (driving pressure ≥ 15mbar) are reached, then the advisory displays a recommendation to rethink the patient's ventilation strategy. Furthermore, permissive hypercapnia and oxygen saturating limits considered as safe will be given. (paCO2: 55mmHg, pH: 7.25, paO2: 80 mmHg, SaO2: 92%)

DETAILED DESCRIPTION:
Background Lung protective ventilation is a well-established treatment to reduce ventilator-induced lung injury (VILI) in patients suffering from ARDS. To quantify lung protective ventilation the concept of driving pressure (ΔP) and mechanical power were postulated.

Although low tidal volumes and low driving pressures are considered standard of care, it was shown that lung protective ventilation is very little used in ICU patients. Especially in those with a less severe lung disease.

Automated Clinical Decision Support (CDS) systems are gaining more attention in clinical practice. They have been successfully used to increase medical provider adherence to guidelines or local department policy. Another successful means of influencing behavior of medical providers are so called nudge-based interventions. Currently there is little evidence on nudge-type interventions or automated alerts for ventilator settings in the ICU. To our knowledge studies that linked these interventions to a change in patient's outcome are lacking.

Hypothesis Activation of an advisory in the patient data management system accompanied by educational sessions and feedback emails decrease ventilation driving pressure in mechanically ventilated patients at increased risk of ARDS (LIPS ≥ 4). As secondary outcome parameters, incidence of ARDS, ventilator free days, reintubation rate, length of stay in the ICU or the hospital and mortality at day 28 will be evaluated.

Methods As an advisory is activated in the ICU software, medical staff caring for the patients can't be blinded. Therefore, the trial will be conducted as observational cohort trial. During the first six month all patients with a LIPS ≥ 4 will be included in the control group. No change of care is needed. In a second phase during the next six months, all patients with a LIPS ≥ 4 will be included into the alert group where advisories will be shown in the patient data management system.

To create this advisory, a clinical advisory rule is executed every 4 hours and the appropriate advisory text is calculated. If the defined threshold values (driving pressure ≥ 15mbar) are reached, then the advisory displays a recommendation to rethink the patient's ventilation strategy. Furthermore, permissive hypercapnia and oxygen saturating limits considered as safe will be given. (paCO2: 55mmHg, pH: 7.25, paO2: 80 mmHg, SaO2: 92%)

Outcome The primary outcome is an improvement of medical stuff's adherence to current recommendations shown by a reduction of the mean ventilator driving pressure (by using the AUC of driving pressures).

The secondary outcomes are ventilator free days, 28-day mortality, reintubation rate, incidence of ARDS and length of stay in the ICU and the hospital.

ELIGIBILITY:
Inclusion Criteria:

* LIPS >= 4, ventilated invasively at point of screening

Exclusion Criteria:

* ARDS at admission
* Pregnant patients
* Age < 18 years
* Patients with elevated intracranial pressure

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at risk of ARDS at six intensive care units will be included in this trial. Study population will consist of medical and surgical ICU patients.
Sampling Method: Non-Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Change of AUC of driving pressure | 10 days
  The driving pressure will be used to create a graph; The AUC will be calculated for each patient. Changes in AUC will be used as measurement for driving pressure over time.

SECONDARY OUTCOMES:
Change in ventilator free days | Day 1-28
28-day mortality, 90-day mortality and one-year mortality | 1 Year
Change in ARDS incidence | Day 1-28
Reintubation rate due to respiratory failure | Day 1-28
Reduction of mechanical power | Day 1-10

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No